CLINICAL TRIAL: NCT03856125
Title: Effectiveness of a Combined Treatment Percutaneous Electrical Stimulation on Radial Nerve With an Exercise Program in Patients With Lateral Epicondylalgia
Brief Title: Percutaneous Electrical Stimulation on Radial Nerve in Patients With Lateral Epicondylalgia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid19 locked down
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CI: 19/043
Record Dates: First submitted 2019-02-20; First posted 2019-02-27 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Lateral Epicondylitis
Keywords: Tennis elbow; Lateral epicondylalgia; Lateral elbow tendinopathy; Lateral elbow pain; Percutaneous electrical stimulation
MeSH Terms: conditions — Tennis Elbow | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENS plus exercise group (Experimental): 4-week intervention program with 2 weekly treatment sessions, one of percutaneous electrical stimulation and supervised exercise and the other one, domiciliary exercise.
  Interventions: Other: PENS plus exercise
- Sham PENS plus exercise group (Sham Comparator): 4-week intervention program with 2 weekly treatment sessions, one of sham percutaneous electrical stimulation and supervised exercise and the other one, domiciliary exercise.
  Interventions: Other: Sham PENS plus exercise

INTERVENTIONS:
Other: PENS plus exercise — The technique will be performed ultrasound-guided on the radial nerve, the places of the needle's insertions will be the following:
  * Needle will be placed at under the lateral intermuscular septum between the triceps brachii and brachialis, approximately 10cm superior to the lateral epicondyle
  * Needle will be placed at the upper third of the forearm on the posterior interosseous nerve after passing the arcade of Froshe's
  The percutaneous electrical stimulation will be realized with a transcutaneous electric nerve stimulation (TENS) current:
  * TENS Frequency - 2 Hz
  * TENS Pulse width - 250 microseconds
  * Duration - 30 minutes.
  * TENS Intensity - Increased at an intensity of visible motor response of the innervated musculature and maximal tolerable intensity.
  * Administration - One per week
  Arms: PENS plus exercise group
Other: Sham PENS plus exercise — The technique will be performed on the radial nerve, the places of the needle's. The technique will be performed ultrasound-guided on the radial nerve, the places of the needle's insertions will be the following:
  * Needle will be placed at under the lateral intermuscular septum between the triceps brachii and brachialis, approximately 10cm superior to the lateral epicondyle.
  * Needle wil be placed at the at the upper third of the forearm on the posterior interosseous nerve after passing the arcade of Froshe's.
  The current will not be working, and the needles will be placed during 30 minutes.
  - Administration - One per week
  Arms: Sham PENS plus exercise group

SUMMARY:
Lateral epicondylalgia is a common musculoskeletal condition that approximately affects 1-3% of the general population. Several authors have found greater mechanical pain sensitivity in the radial nerve when compared with healthy subjects. Radial tunnel syndrome exhibits a similar clinical presentation to lateral epicondylalgia. Percutaneous electrical stimulation has shown reduce pain in several conditions. Percutaneous electrical stimulation on the radial nerve could cause an important relief in lateral epicondylalgia.

Hypothesis: Percutaneous electrical stimulation on radial nerve plus exercise therapy in patients with lateral epicondylalgia is better than sham percutaneous electrical stimulation plus exercise.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo controlled clinical trial, using Percutaneous Electrical Nerve Stimulation (PENS). PENS is technique to provide a transcutaneous electrical nerve stimulation current throughout needling filaments place close to the nerve.

Study Aims:

Aim #1: The primary aim of the study is to compare the effect of the immediate, short, medium and long-term of PENS on intensity of pain as measured by visual analogue scale (VAS) in patients with lateral epicondylalgia with random assignment to two treatments: PENS plus exercise program or Sham PENS plus exercise program.

Aim #2: The secondary aim of the study is to compare the effect of the immediate, short, medium and long-term of PENS on pain free grip strength, disability as measured by Patient Rated Tennis Elbow Evaluation (PRTEE) and DASH questionnaire and pressure pain threshold (PPT) and area and distribution of pain in patients with lateral epicondylalgia with random assignment to two treatments: PENS plus exercise program or Sham PENS plus exercise program, and determine if psychological factors (fear and avoidance and catastrophism) change with any of the treatments and if is related with the primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Lateral epicondylalgia symptoms confirmed with at least 2 of the 4 following test:

  1. pain during palpation of lateral epicondyle
  2. pain on resisted wrist extension
  3. pain on resisted middle finger extension
  4. pain during hand-grip.

Exclusion Criteria:

* History of fractures, luxations, surgery and/or musculoskeletal disorders in upper limb.
* Neurological disorders, inflammatory and/or degenerative diseases.
* Having received as treatment techniques that involve needles on the previous 6 months to study enrollment, or having received percutaneous electrical stimulation as a treatment before.
* Cervical pathology, fibromyalgia, unstable cardiovascular diseases, pregnant women or under suspect of pregnancy.
* Contraindications of needle's insertions: anticoagulant therapy, needle phobia, diabetes, hypothyroidism, lymphoedema, muscular diseases).
* Contraindications of electrical current application.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-05-21 (Actual)

PRIMARY OUTCOMES:
Pain Intensity: visual analogue scale | Change from baseline to immediate (single session); 4 weeks; 8 weeks; 16 weeks; 28 weeks; 52 weeks
  Pain intensity measured with a 100mm (0 - No pain - 100 The worst pain) visual analogue scale

SECONDARY OUTCOMES:
Patient Rated Tennis Elbow Evaluation (PRTEE) | Change from baseline to 4 weeks; 8 weeks; 16 weeks; 28 weeks; 52 weeks
  It is a 15-item questionnaire designed to measure forearm pain and disability in patients with lateral epicondylitis. The PRTEE allows patients to rate their levels of tennis elbow pain and disability from 0 to 10, and consists of 2 subscales: pain and function.
Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire | Change from baseline to 4 weeks; 8 weeks; 16 weeks; 28 weeks; 52 weeks
  It includes 30 items assessing (1) degree of difficulty during the preceding week in performing several physical activities because of problems in a upper extremity (21 items), (2) severity of each of the symptoms of pain, activity-related pain, tingling, weakness, and stiffness (5 items), and (3) the problem's effect on social activities, work, and sleep and its psychological impact (4 items). Each item is answered on a 5-point scale ranging from 1 (no difficulty to perform, no symptom, or no impact) to 5 (unable to do, very severe symptom, or high impact). The responses to the 30 items are summed to form a raw score that is then converted to a scale from 0 to 100 with a formula. A higher score reflects greater disability.
Pain free grip strength | Change from baseline to immediate (single session); 4 weeks; 8 weeks; 16 weeks; 28 weeks
  Measurement the amount of force that the patient generates to the onset of pain as measured with a dynamometer
Pressure pain threshold using an algometer | Change from baseline to immediate (single session); 4 weeks; 8 weeks; 16 weeks; 28 weeks; 52 weeks
  Measurement of pressure pain threshold in the lateral epicondyle, radial nerve in the spiral groove, C5-C6 zygapophyseal joints, and the tibialis anterior muscle.
Area of pain | Change from baseline to 4 weeks; 8 weeks; 16 weeks; 28 weeks; 52 weeks
  The participants will paint the area of extension of their pain in a body chart. The area in mm^2 will be calculated using a software
Pain distribution | Change from baseline to 4 weeks; 8 weeks; 16 weeks; 28 weeks; 52 weeks
  The pain distribution will be classified as 0=no pain, 1=pain only proximal and lateral elbow, 2=distal pain to the elbow (forearm and wrist), 3= pain in other regions (arm, shoulder and neck) using the painted region in the body chart
Kinesiophobia | Change from baseline to 4 weeks; 8 weeks; 16 weeks; 28 weeks; 52 weeks
  Tampa Scale for Kinesiophobia. To assess the fear of movement and pain-related fear. The 11 items are scored 1-4, with total scores ranging from 11 to 44. The addition of all the points obtained from each of the items results in the level of kinesiophobia, with higher scores indicating greater perceived kinesiophobia
Pain catastrophizing | Change from baseline to 4 weeks; 8 weeks; 16 weeks; 28 weeks; 52 weeks
  Pain Catastrophizing Scale (PCS). This tool is a 13-item questionnaire designed to measure the three components of pain-related catastrophizing: rumination, magnification, and helplessness, resulting in a unique score. Each item is responded to on a 5-point scale (0 not at all, 4 all the time) relating the degree to which the individual experiences a thought or feeling of a painful situation.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Complutense de Madrid, Madrid, Spain